CLINICAL TRIAL: NCT07111975
Title: ANEURYSM@RISK: Automatic Intracranial Aneurysm Quantification and Feature Learning Modelling to Optimize Intracranial Aneurysm Rupture Prediction
Status: Active, not recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Bichat Hospital (Other); University Medical Center Hamburg-Eppendorf (UKE) (Unknown); Philips Medical Systems (Industry)
Responsible Party: Principal Investigator, Phebe J Groenheide, MSc, PhD Candidate, Department of Radiology/Neurology, UMC Utrecht
Other Study IDs: 23U-0036_AWARE
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Aneurysms; Unruptured Intracranial Aneurysm; Subarachnoid Hemorrhage (SAH) From Ruptured Aneurysm
Keywords: Artificial Intelligence; Intracranial Aneurysm; Brain Aneurysm; Unruptured Intracranial Aneurysm; MR Angiography; 3D Segmentation; Rupture/Growth Risk Prediction; Subarachnoid Hemorrhage; Clinical Decision Support; SHERPA; UMC Utrecht; Morphology; Shape
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stable Intracranial Aneurysm Group: Participants with unruptured intracranial aneurysms (UIAs) that remained stable over time, showing no morphological growth or rupture during follow-up. Data are sourced from UMC Utrecht, UKE Hamburg, and AP-HP Paris.
- Unstable Intracranial Aneurysm Group: Participants with intracranial aneurysms (IAs) that demonstrated instability over time, defined as morphological growth and/or rupture during follow-up. Data are sourced from UMC Utrecht, UKE Hamburg, and AP-HP Paris.

SUMMARY:
ANEURYSM@RISK is an observational study aiming to develop and validate an artificial intelligence (AI)-based prediction model for the growth and rupture of intracranial aneurysms (IAs). By applying automated 3D segmentation and morphological quantification of IAs from MR angiography (MRA) scans, the model is intended to provide clinicians with objective and reproducible risk estimates of aneurysm instability.

The study utilizes retrospective imaging data from multiple European centers, including UMC Utrecht, AP-HP Paris, and University Medical Center Hamburg-Eppendorf (UKE). A clinical vignette study will evaluate the model's clinical utility and user experience among interventional radiologists.

This study is exempt from medical ethics review (non-WMO in the Netherlands), as it involves only existing, anonymized data and imposes no additional burden on patients.

DETAILED DESCRIPTION:
The ANEURYSM@RISK study is part of the SHERPA project (Smart Human-centred Effortless support for Professional clinical Applications). The study aims to develop and validate a multivariable artificial intelligence (AI)-based prediction model to identify unstable unruptured intracranial aneurysms (UIAs), using morphological and clinical features.

Retrospective MR angiography (MRA) data will be collected from three clinical sites: UMC Utrecht (The Netherlands), AP-HP Paris (France), and University Medical Center Hamburg-Eppendorf (Germany). The study workflow includes:

* Development of AI algorithms for 3D shape feature extraction after automated aneurysm segmentation
* Training of predictive models for aneurysm growth and rupture based on morphological and clinical parameters
* Validation of model performance using a longitudinal dataset of ~1,000 patients (target C-statistic ≥ 0.80)
* A clinical vignette study in real-life settings to evaluate usability, decision-making impact, and inter-clinician variability

Key Performance Indicators (KPIs):

* Discriminative performance for aneurysm instability prediction; C-statistic ≥ 0.80
* Sensitivity ≥ 80% and specificity ≥ 50% (based on optimal cut-off values)
* ≥ 25% reduction in time to clinical decision-making
* ≥ 80% adherence to AI-generated suggestions by interventional radiologists
* ≥ 20% improvement in user experience using 3D visualization compared to 2D displays (survey-based)
* ≥ 50% reduction in inter- and intra-observer variability in aneurysm assessment

Ethical Considerations:

This is a non-interventional, retrospective study using previously acquired and anonymized imaging data. No additional procedures or data collection will be performed. The study poses no added burden or risk to patients. According to Dutch regulations, it is not subject to the Medical Research Involving Human Subjects Act (non-WMO).

ELIGIBILITY:
Inclusion Criteria:

* Available MR angiography (MRA) scans of the Circle of Willis
* Presence of at least one intracranial aneurysm (IA)
* Availability of follow-up imaging or clinical records indicating stability, growth, or rupture

Exclusion Criteria:

* Imaging of insufficient quality for segmentation or analysis
* Lack of follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosed unruptured intracranial aneurysms (UIAs) identified through MR angiography imaging, with follow-up records, from three European academic hospitals. All data are retrospective and anonymized.
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Discriminative performance of AI model for aneurysm instability prediction | At time of model validation; Up to 36 months from study start
  Model performance measured by C-statistic (AUC) with a target threshold of ≥ 0.80. Instability is defined as aneurysm growth and/or rupture during follow-up.

SECONDARY OUTCOMES:
Sensitivity and specificity of AI model | At time of model validation; Up to 36 months from study start
  Targets: Sensitivity ≥ 80% and specificity ≥ 50%, based on optimal cut-off derived from ROC analysis.
Reduction in inter- and intra-observer variability | During vignette study in clinical setting; During final 6 months of study
  Measured as reduction in variation in risk classification between and within clinicians. Target: ≥ 50% reduction.
Clinician adherence to AI suggestions | During vignette study; During final 6 months of study
  Proportion of cases where interventional radiologists follow AI risk estimates in their decision-making. Target adherence: ≥ 80%.
Reduction in clinical decision-making time | During vignette study; During final 6 months of study
  Time required for clinical decision-making with AI compared to without AI. Target reduction: ≥ 25%.
User satisfaction with AI tool | Immediately after using the AI tool in vignette study; During final 6 months of study
  Self-reported satisfaction measured using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied). Higher scores indicate greater satisfaction. Target: average score ≥ 4.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center (UMC) Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data derived from imaging, including intracranial aneurysm morphological measurements and risk predictions, will be shared upon reasonable request from qualified investigators.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The individual participant data (IPD) and supporting documentation will be available after the publication of the main study results. The end date for availability has not yet been determined.
Access Criteria: Only qualified academic researchers may request access for non-commercial purposes. Requests must include a description of the intended use and can be directed to: p.j.groenheide@umcutrecht.nl.

REFERENCES:
- See also: SHERPA: Smart Human-centred Effortless support for Professional clinical Applications — https://doi.org/10.3030/101194744
- See also: SHERPA: Smart Human-centred Effortless support for Professional clinical Applications — https://sherpa-ihi.eu/